CLINICAL TRIAL: NCT02269124
Title: Use of Amplification in Children With Unilateral Hearing Loss
Acronym: UHL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Michael Cohen, Principal Investigator, Massachusetts Eye and Ear Infirmary
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2019P000948; 14-006H (Other: Mass Eye and Ear IRB (Obsolete))
Record Dates: First submitted 2014-10-16; First posted 2014-10-20 (Estimated); Results first posted 2021-08-11 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-07

CONDITIONS: Unilateral Hearing Loss
MeSH Terms: conditions — Hearing Loss, Unilateral | interventions — Hearing Aids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional Measures Only (No Intervention): In arm 1, the child will utilize conventional measures for management of unilateral hearing loss, such as FM system and preferential seating in the classroom. While two basic types of FM systems exist, personal and sound field, subjects in our study will utilize a personal FM system, worn at the ear-level. This will increase the likelihood that the child will receive amplification in all classes, and will help to standardize this intervention. The HEAR-QL, CHILD (child) questionnaire, and LIFE-R student questionnaire will be administered to the child at the beginning, midpoint, and conclusion of this 3-month arm via Redcap. The CHILD (parent) questionnaire will be administered to the parent and the LIFE-R teacher questionnaire will be administered to the teacher at the same intervals.
- Conventional Measures + Hearing Aid (Experimental): In arm 2, the child will use the conventional measures described above in addition to a digital behind-the-ear hearing aid with a standard ear hook and custom ear mold on the affected ear. The hearing instrument will be customized by an audiologist. The subject will be instructed to wear the hearing aid both at home and at school. In both arms, the FM system will be used in school only. As in the first arm, the HEAR-QL, CHILD (child) questionnaire, and LIFE-R student questionnaire will be administered to the child at the beginning, midpoint, and conclusion of this 3-month arm. The CHILD (parent) questionnaire will be administered to the parent and the LIFE-R teacher questionnaire will be administered to the teacher at the same intervals. No washout period will take place between the two arms. Subjects will be randomized to complete one arm first for 3 months, followed immediately by 3 months in the opposite arm.
  Interventions: Device: Hearing aid

INTERVENTIONS:
Device: Hearing aid — The subject will wear a hearing aid at all times for a 3-month period. At school, he/she will wear this hearing aid in addition to using conventional measures (FM system and preferential seating).
  Arms: Conventional Measures + Hearing Aid

SUMMARY:
Unilateral hearing loss (UHL) in children has been demonstrated to have a negative impact on quality of life, school performance and behavior. Despite this knowledge, it remains unclear how to best manage this common problem. There has been much debate regarding this issue with many programs recommending preferential seating in the classroom and use of a frequency-modulated (FM) system to amplify the teacher's voice in the classroom (conventional measures), and others recommending these accommodations in addition to use of a hearing aid for amplification (amplification). There is very limited research to support or refute the efficacy of a hearing aid in improving measurable academic, behavioral, or quality-of-life (QOL) outcomes in children with UHL. We propose a study evaluating the impact of hearing aid use in school-aged children (ages 6-12 years) with mild to moderately severe UHL. In this study, subjects will be randomized to receive either conventional measures or conventional measures plus amplification. After a three month period, the groups will be reversed, with each subject serving as their own control. Outcome measurements will include patient reported disease-specific QOL reported by patients, parents, and teachers using validated survey instruments at regular intervals throughout the study period.

DETAILED DESCRIPTION:
Unilateral hearing loss (UHL) is defined as decreased hearing in one ear, with normal hearing thresholds in the contralateral ear. Approximately 0.83/1000 newborn children are found to have UHL. It is estimated that about 3-5% of all children in the United States are eventually diagnosed with UHL. When the cutoff for normal hearing is placed at 15 decibels (dB), this incidence is as high as 6.3%, which corresponds to a prevalence of 6.2 million children nationally. The management of UHL continues to be an area of debate, as the handicap associated with UHL is often underestimated. In fact, those with UHL often go without assistance due to lack of recognition of the disability by some health and educational professionals, who have claimed that this hearing loss "attracts little attention from either patient or parent" and that "these children experience few communicational or educational problems." However, in evaluation of children with permanent hearing loss, rates of children who need speech/language intervention and aural rehabilitation are not significantly different between those with bilateral permanent hearing loss and those with unilateral permanent hearing loss. Unfortunately, children with UHL are half as likely to be referred for hearing testing as those with bilateral hearing loss.

Studies have demonstrated the negative impact of unilateral hearing impairment in children. Educational and behavioral difficulties have been clearly shown, with a number of studies demonstrating increased rates of failure of at least one grade in children with UHL when compared to their classmates with normal hearing (24-35% vs. 3.5%). Additionally, increase in special educational needs (12-41%) and frequent problems with behavior have also been noted in this population. In several studies, Lieu and colleagues have shown poorer performance for children with UHL. In a study looking at oral and written language scores, children with UHL did significantly worse than their siblings, who served as matched controls, on language comprehension, oral expression, and oral composite scores. In addition, these children were four times more likely to have Individualized Education Plans (IEPs) and twice as likely to have received speech-language therapy.

Despite these findings regarding the impact of UHL on children, there is a paucity of literature to support or refute the efficacy of hearing aid use in improving measurable academic, behavioral, or quality-of-life (QOL) outcomes. While hearing related disease-specific quality of life measures for children were not developed until very recently, previous studies in adults with UHL reported decreased quality of life, with increased frustration and shame due to hearing disability. The Hearing Environments and Reflection on Quality of Life questionnaire, or HEAR-QL, an instrument developed and validated at Washington University in St. Louis for young children with hearing loss initially (2011) and then later for adolescents (2013), examined effects on environments, activities, and feelings of children with both unilateral and bilateral hearing loss. Significantly lower scores, indicating poorer quality of life, were seen in patients with both UHL and bilateral hearing loss. Interestingly, differences in quality of life between children with UHL and children with bilateral hearing loss were found to be significant in only 1 out of 3 subdomains.

A 2010 study by Johnstone et al. demonstrated that children with UHL who used amplification at a young age (6-9 years) had improvement in localization acuity, while those who received amplification at an older age (10-14 years) noted impairment in localization. This may indicate that the timing of initiation of amplification in UHL may play an important role in whether the intervention is beneficial. In addition, Noh and Park's study in 2012 demonstrated that children with UHL needed to sit 3.5 meters closer to the teacher to obtain the same speech discrimination scores as children with binaural hearing. While this can be accomplished in a small room setting, this may not be possible at all times in all classes, and it is certainly not translatable to hearing environments outside of the classroom. It is not clear whether adding amplification to would eliminate this handicap and improve quality of life, behavior, or academic performance.

Current interventions: Multiple options exist for management of UHL. Preferential seating in the classroom is often the first line of treatment utilized, placing the child at the front of the classroom with the better hearing ear toward the teacher. Evaluation of the classroom by an educational audiologist or other specialist in the education of children with hearing loss in order to optimize the listening environment is another commonly utilized modality for managing UHL. Interventions such as carpeting, tennis balls placed on the legs of chairs, and selection of a classroom with lower ambient noise levels from outside traffic or air handling equipment can reduce significantly improve signal to noise ratios for the student. Another modality for improving signal to noise ration is use of a frequency-modulated (FM) system in the classroom, which specifically amplifies the teacher's voice via a microphone worn by the teacher. This increases the signal-to-noise ratio for the teacher's voice as it does not amplify background noise. Differentiating relevant sound signals from background noise a particularly challenging problem for children with UHL. Other options for management of UHL include various forms of amplification including a unilateral hearing aid, contralateral routing of sound (CROS) systems, and potentially cochlear implantation (though this practice has not been widely adopted in children with UHL in the United States).

In the only study to date comparing the above modalities to one another, Updike compared speech perception measures in 6 children, ages 5 to 12 years, with mild to profound UHL with use of FM systems, CROS aids, and conventional hearing aids. He concluded that FM systems were beneficial in all hearing situations and in all degrees of hearing loss. In addition, he stated that neither hearing aids nor CROS aids provided benefit in speech understanding, and both may worsen speech perception in noisy situations. Multiple limitations exist with this study, including a small sample size and lack of a time period for the patients to adjust to the use of amplification.

In studies looking at acceptance of hearing aid use in children with UHL, children with mild to moderately severe hearing loss tended to accept hearing aids, while those with severe to profound hearing loss were less accepting. Parental satisfaction with hearing aids in this population has been good, with many noticing improved hearing for their children. More recently, Briggs et al. published a study looking at 8 children, ages 7 to 12 years, with mild to moderately severe UHL, who were aided with digital hearing aids. Although speech perception scores did not show significant improvement, parents subjectively reported significant improvement in quality of life after 3 months of use. In one German study of 3 children with severe to profound unilateral hearing loss, improvement in speech understanding in noise and sound localization following cochlear implantation was observed and subjective improvement was reported by parents.

Compliance with use of amplification should also be considered in these cases, as Fitzpatrick et al. demonstrated in a study of 670 children with unilateral or bilateral hearing loss. While amplification was recommended in 90%, less than two-thirds of the children wore their hearing aids consistently.

To date, only two studies exist which examine the use of amplification in children with unilateral hearing loss. Both studies are limited by small sample size. In addition, the earlier study evaluated analog hearing aids, whereas in the present day, digital hearing aids are widely used, and was further limited by a very short study period. Our study proposes to examine whether children with UHL note improved quality of life when using amplification via a hearing aid in conjunction with conventional classroom accommodations including an FM system.

In our study we will compare the use of conventional measures to conventional measures plus a digital hearing aid on the affected ear using validated quality of life instruments administered to the subject, the subject's teacher, and the subject's parent. The instruments used will be the HEAR-QL, the CHILD, and the LIFE-R (See outcome measures for details).

Each of the surveys will be administered five times in total: at the time of enrollment, once at the midpoint of the first treatment arm, once after completion of the first treatment arm, once at the midpoint of the second treatment arm, and once after completion of the second treatment arm. Comparisons will then be made among groups as described later in this proposal.

Our practice is well suited to carrying out this study as we are a tertiary care center serving a large region. Our multidisciplinary pediatric hearing loss clinic allows children to be evaluated and longitudinally followed in conjunction with the audiology, speech and language pathology, neuropsychology, and medical genetics. In the past year, there were over 300 visits coded for unilateral hearing loss based on ICD-9 codes, with 70 unique patients, making recruitment of our target sample size over the 3-year study period feasible. The potential impact of this study is great, as there is no consensus as to whether amplification should be recommended for children with unilateral hearing loss, and a study of this power would serve as a useful guide in this decision-making process.

ELIGIBILITY:
Inclusion Criteria:

Children ages 6-12 years with mild to moderately severe unilateral hearing loss, with thresholds across 4 frequencies ≥ 25 dB but < 70 dB in the worse hearing ear; Normal hearing in the contralateral ear, defined as thresholds ≤ 20 dB from 250 Hz to 8000 Hz; Unaided word recognition scores of ≥ 80% in worse hearing ear

Exclusion Criteria:

Contralateral hearing loss; Significant cognitive impairment; Middle ear disease that has not been addressed; Inability to commit to treatment program

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Cohen, MD, Principal Investigator — Massachusetts Eye and Ear Infirmary
Locations (1):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Benchetrit L, Stenerson M, Ronner EA, Leonard HJ, Aungst H, Stiles DJ, Levesque PA, Kenna MA, Anne S, Cohen MS. Hearing Aid Use in Children With Unilateral Hearing Loss: A Randomized Crossover Clinical Trial. Laryngoscope. 2022 Apr;132(4):881-888. doi: 10.1002/lary.29829. Epub 2021 Aug 20. PMID 34415079

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 442 children were assessed for eligibility based on presence of mild to moderately-severe UHL and > 80% word recognition scores. Of these, 325 did not meet eligibility criteria and 80 declined to participate. Thirty-seven children were enrolled from Massachusetts Eye and Ear (n=25), Boston Children's Hospital (n=5), and Cleveland Clinic (n=7) between 2014 and 2019. Thirty-four children completed study interventions. There was no washout period between arms.
Groups:
- Conventional Measures Only First; Then Conventional Measures + Hearing Aid: This group was randomized to complete the 3-month "Conventional Measures Only" arm first, followed immediately by the 3-month "Conventional Measures + Hearing Aid" arm. There was no washout period between arms.
- Conventional Measures + Hearing Aid First; Then Conventional Measures Only: This group was randomized to complete the 3-month "Conventional Measures + Hearing Aid" arm first, followed immediately by the 3-month "Conventional Measures Only" arm. There was no washout period between arms.
Period: Overall Study
Arm/Group | Conventional Measures Only First; Then Conventional Measures + Hearing Aid | Conventional Measures + Hearing Aid First; Then Conventional Measures Only
Started (Completion of each of the six survey rounds is defined here as completing at least one of the five surveys for the given time point.) | 21 | 16
Completed Survey Round 1 (Arm 1, 0 Weeks) (Survey Round 1 was administered 0 weeks into the study, corresponding to the beginning of the first treatment arm. Round 1 represents the first of six survey rounds overall.) | 20 | 14
Completed Survey Round 2 (Arm 1, 6 Weeks) (Survey Round 2 was administered 6 weeks into the study, corresponding to the halfway point within the first treatment arm. Round 2 represents the second of six survey rounds overall.) | 17 | 13
Completed Survey Round 3 (Arm 1, 12 Weeks) (Survey Round 3 was administered 12 weeks into the study, corresponding to the last measures during the first treatment arm. Survey Round 3 was administered shortly before the subject had ended the first treatment arm, while Survey Round 4 was administered shortly after the subject initiated the second treatment arm. Round 3 represents the third of six survey rounds overall.) | 17 | 11
Completed Survey Round 4 (Arm 2, 12 Weeks) (Survey Round 4 was administered 12 weeks into the study, corresponding to the first measures during the second treatment arm. Survey Round 4 was administered shortly after the subject had initiated the second treatment arm, while Survey Round 3 was administered shortly before the subject ended the first treatment arm. Round 4 represents the fourth of six survey rounds overall.) | 11 | 8
Completed Survey Round 5 (Arm 2, 18 Weeks) (Survey Round 5 was administered 18 weeks into the study, corresponding to the halfway point within the second treatment arm. Round 5 represents the fifth of six survey rounds overall.) | 16 | 10
Completed Survey Round 6 (Arm 2, 24 Weeks) (Survey Round 6 was administered 24 weeks into the study, corresponding to the last measures in the second treatment arm. Round 6 represents the sixth of six survey rounds overall.) | 14 | 10
Completed (Overall completion is defined here as completing at least one survey.) | 20 (One participant from the Conventional Measures Only First arm did not return any surveys, nor did their parent/guardian or teacher, and were deemed lost to follow-up.) | 14 (Two participants from the Conventional measures + Hearing Aid First arm withdrew from the study prior to the second arm because they did not wish to stop using the hearing aid.)
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Conventional Measures Only First, Then Conventional Methods + Hearing Aid: Of the participants who completed the study, twenty (20) were assigned to complete the 3-month "Conventional Measures Only" arm first, during which only FM system and preferential seating were used. After this first 3-month arm, these participants then immediately proceeded to complete the second 3-month "Conventional Measures + Hearing Aid" arm, during which conventional measures and a hearing aid was used.
- Conventional Measures + Hearing Aid First, Then Conventional Methods Only: Of the participants who completed the study, fourteen (14) were assigned to complete the 3-month "Conventional Measures + Hearing Aid" arm first, during which an FM system, preferential seating, and a hearing aid were all used. After this first 3-month arm, these participants then immediately proceeded to complete the second 3-month "Conventional Measures Only" arm, during which only FM system and preferential seating were used.
- Total: Total of all reporting groups
Arm/Group | Conventional Measures Only First, Then Conventional Methods + Hearing Aid | Conventional Measures + Hearing Aid First, Then Conventional Methods Only | Total
Number analyzed (Participants) | 20 | 14 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 14 | 34
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.9 (1.5) | 8.1 (1.6) | 8.0 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 21
  Male | 8 | 5 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 18 | 11 | 29
  Black | 0 | 2 | 2
  Other/Unknown | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 14 | 34
Hearing loss severity [Count of Participants; unit: Participants]
  Mild-moderate (20-60 dB PTA) | 17 | 11 | 28
  Moderate-severe (60-75 dB PTA) | 3 | 3 | 6
Hearing loss type [Count of Participants; unit: Participants]
  Conductive | 13 | 7 | 20
  Sensorineural | 7 | 6 | 13
  Mixed | 0 | 1 | 1
Hearing loss progression [Count of Participants; unit: Participants]
  Stable | 15 | 13 | 28
  Fluctuating | 4 | 0 | 4
  Progressive | 1 | 1 | 2
Hearing loss etiology [Count of Participants; unit: Participants]
  Congenital | 7 | 3 | 10
  Acquired | 13 | 8 | 21
  Unknown | 0 | 3 | 3
FM system use prior to trial entry [Count of Participants; unit: Participants]
  Yes | 12 | 9 | 21
  No | 7 | 5 | 12
  Unknown | 1 | 0 | 1
State and Hospital of Enrollment [Count of Participants; unit: Participants]
  Massachusetts (Massachusetts Eye and Ear) | 14 | 9 | 23
  Massachusetts (Boston Children's Hospital) | 2 | 2 | 4
  Massachusetts Total | 16 | 11 | 27
  Ohio (Cleveland Clinic) | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: HEAR-QL 26 Questionnaire
Description: The HEAR-QL consists of 28 items that measure the perceived effect of hearing loss on quality of life. It is adjusted to a scale of 0-100, with lower scores indicating a worse disease-specific quality of life and higher scores signifying a better disease-specific quality of life. The HEAER-QL-26 was one of three surveys used to evaluate the study's primary endpoint: subject-reported quality of life.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Conventional Methods Only First, Then Conventional Methods + Hearing Aid: Subjects randomized into the "conventional methods arm" began participating in the study using only conventional methods (FM system and preferential seating in school). Subjects used conventional methods only for 3 months, followed by 3 months using all conventional methods plus a hearing aid. Presented here are averages and standard deviations of survey scores completed by participants randomized into this group at each of the 6 time points, with rounds 1-3 representing conventional methods only and rounds 4-6 representing conventional methods with a hearing aid.
- Conventional Methods + Hearing Aid First, Then Conventional Methods Only: Subjects randomized into the "conventional methods + hearing aid arm" began participating in the study using all conventional methods (FM system and preferential seating in school) in addition to a hearing aid. Subjects used a hearing aid along with all conventional methods for 3 months, followed by 3 months using conventional methods only. Presented here are averages and standard deviations of survey scores completed by participants randomized into this group at each of the 6 time points, with rounds 1-3 representing conventional methods with a hearing aid and rounds 4-6 representing conventional methods only.
Arm/Group | Conventional Methods Only First, Then Conventional Methods + Hearing Aid | Conventional Methods + Hearing Aid First, Then Conventional Methods Only
Number analyzed (Participants) | 20 | 14
score on a scale
  Survey Round 1 (Arm 1, 0 Weeks) | 69.61 (15.06) | 74.05 (15.14)
  Survey Round 2 (Arm 1, 6 Weeks) | 71.04 (18.29) | 80.21 (16.22)
  Survey Round 3 (Arm 1, 12 Weeks) | 74.31 (20.43) | 87.15 (10.48)
  Survey Round 4 (Arm 2, 12 Weeks) | 77.78 (26.06) | 76.31 (22.86)
  Survey Round 5 (Arm 2, 18 Weeks) | 79.13 (21.75) | 73.32 (24.32)
  Survey Round 6 (Arm 2, 24 Weeks) | 80.42 (23.14) | 75.17 (23.03)

2. Primary Outcome: CHILD (Child) Questionnaires
Description: The CHILD (child) questionnaire consists of 15 questions that describe situations where hearing difficulty may occur when the child is with his/her family. The answers are measured on a scale of 1-8, with 1 indicating poor ability to hear, and 8 indicating complete understanding. The total scores across all questions were standardized on a scale of 0 to 100, with lower scores indicating a worse disease-specific quality of life and higher scores signifying a better disease-specific quality of life. Two versions, the CHILD (child) and the CHILD (parent) are phrased to apply to the child and the parent respectively. The CHILD (child) was one of three surveys used to evaluate the study's primary endpoint: subject-reported quality of life.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Conventional Methods Only First, Then Conventional Methods + Hearing Aid | Conventional Methods + Hearing Aid First, Then Conventional Methods Only
Number analyzed (Participants) | 20 | 14
score on a scale
  Survey Round 1 (Arm 1, 0 Weeks) | 69.21 (21.55) | 72.83 (16.51)
  Survey Round 2 (Arm 1, 6 Weeks) | 75.23 (17.28) | 82.83 (9.64)
  Survey Round 3 (Arm 1, 12 Weeks) | 77.59 (13.78) | 80.13 (14.18)
  Survey Round 4 (Arm 2, 12 Weeks) | 90.36 (10.55) | 67.16 (20.83)
  Survey Round 5 (Arm 2, 18 Weeks) | 81.76 (18.69) | 65.42 (26.41)
  Survey Round 6 (Arm 2, 24 Weeks) | 88.61 (11.83) | 70.43 (23.66)

3. Primary Outcome: LIFE-R Student Questionnaires
Description: The LIFE-R Student questionnaire consists of 15 questions that describe situations where hearing difficulty may occur in school. The answers are measured on a scale of 1-5, with 1 indicating situations in which hearing is always difficult and 5 indicating situations where hearing is always easy. The scores are then added standardized from 0 to 100, with lower scores representing a higher frequency of hearing difficulties in the classroom and higher score representing a lower frequency of hearing difficulties. Two versions, the LIFE-R student and the LIFE-R teacher are phrased to apply to the student and the teacher respectively. The LIFE-R Student questionnaire is one of three surveys used to evaluate the primary endpoint: subject-reported quality of life.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Conventional Methods Only First, Then Conventional Methods + Hearing Aid | Conventional Methods + Hearing Aid First, Then Conventional Methods Only
Number analyzed (Participants) | 20 | 14
score on a scale
  Survey Round 1 (Arm 1, 0 Weeks) | 58.83 (18.86) | 67.05 (15.29)
  Survey Round 2 (Arm 1, 6 Weeks) | 62.81 (19.78) | 77.05 (13.25)
  Survey Round 3 (Arm 1, 12 Weeks) | 64.78 (17.90) | 80.37 (15.18)
  Survey Round 4 (Arm 2, 12 Weeks) | 78.76 (15.15) | 63.13 (23.68)
  Survey Round 5 (Arm 2, 18 Weeks) | 75.94 (18.79) | 62.22 (24.09)
  Survey Round 6 (Arm 2, 24 Weeks) | 80.15 (16.07) | 63.89 (25.00)

4. Secondary Outcome: LIFE-R Teacher
Description: The LIFE-R Teacher questionnaire consists of 14 questions that evaluate the student's academic performance, including ability to focus, follow directions, and understand scholastic material when verbally administered. The answers are measured on a scale of 1-5, with 1 indicating a point of constant challenge for the student and 5 indicating no challenge. The scores are then added and standardized from 0 to 100, with lower scores representing a higher frequency of hearing difficulties in the classroom and higher score representing a lower frequency of hearing difficulties. Two versions, the LIFE-R student and the LIFE-R teacher are phrased to apply to the student and the teacher respectively. The LIFE-R Teacher questionnaire was used to evaluate one of the secondary endpoints: classroom performance.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Conventional Methods Only First, Then Conventional Methods + Hearing Aid | Conventional Methods + Hearing Aid First, Then Conventional Methods Only
Number analyzed (Participants) | 20 | 14
score on a scale
  Survey Round 1 (Arm 1, 0 Weeks) | 68.69 (20.80) | 83.55 (11.00)
  Survey Round 2 (Arm 1, 6 Weeks) | 73.66 (19.55) | 90.61 (6.82)
  Survey Round 3 (Arm 1, 12 Weeks) | 74.26 (17.63) | 89.77 (9.74)
  Survey Round 4 (Arm 2, 12 Weeks) | 75.74 (19.47) | 79.57 (15.54)
  Survey Round 5 (Arm 2, 18 Weeks) | 83.31 (17.81) | 78.08 (19.96)
  Survey Round 6 (Arm 2, 24 Weeks) | 83.94 (16.08) | 83.27 (16.73)

5. Secondary Outcome: CHILD (Parent) Questionnaire
Description: The CHILD (parent) questionnaire consists of 15 questions that describe situations where hearing difficulty may occur when the child is with his/her family. The answers are measured on a scale of 1-8, with 1 indicating poor ability to hear, and 8 indicating complete understanding. The total scores across all questions were standardized on a scale of 0 to 100, with lower scores indicating a worse disease-specific quality of life and higher scores signifying a better disease-specific quality of life. Two versions, the CHILD (child) and the CHILD (parent) are phrased to apply to the child and the parent respectively. The CHILD (parent) survey was used to evaluate one of the study's secondary endpoints: impact of hearing aid with respect to parental perception.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Conventional Methods Only First, Then Conventional Methods + Hearing Aid: Subjects randomized into the "conventional methods arm" began participating in the study using only conventional methods (FM system and preferential seating in school). Subjects used conventional methods only for 3 months, followed by 3 months using all conventional methods and a hearing aid. Presented here are averages and standard deviations of survey scores completed by participants randomized into this group at each of the 6 time points, with rounds 1-3 representing conventional methods only and rounds 4-6 representing conventional methods with a hearing aid.
Arm/Group | Conventional Methods Only First, Then Conventional Methods + Hearing Aid | Conventional Methods + Hearing Aid First, Then Conventional Methods Only
Number analyzed (Participants) | 20 | 14
score on a scale
  Survey Round 1 (Arm 1, 0 Weeks) | 68.52 (19.57) | 73.40 (12.96)
  Survey Round 2 (Arm 1, 6 Weeks) | 67.24 (13.52) | 81.81 (10.29)
  Survey Round 3 (Arm 1, 12 Weeks) | 72.77 (16.70) | 81.73 (12.79)
  Survey Round 4 (Arm 2, 12 Weeks) | 91.24 (5.78) | 64.19 (19.93)
  Survey Round 5 (Arm 2, 18 Weeks) | 85.93 (15.31) | 68.13 (26.41)
  Survey Round 6 (Arm 2, 24 Weeks) | 84.27 (14.47) | 63.10 (23.81)

ADVERSE EVENTS:
Description: All-cause mortality, serious, and other (not including serious) adverse events were not monitored/assessed.
Groups:
- Conventional Measures Only First; Then Conventional Measures + Hearing Aid: This group was randomized to complete the 3-month "Conventional Measures Only" arm first, followed immediately by the 3-month "Conventional Measures + Hearing Aid" arm.
- Conventional Measures + Hearing Aid First; Then Conventional Measures Only: This group was randomized to complete the 3-month "Conventional Measures + Hearing Aid" arm first, followed immediately by the 3-month "Conventional Measures Only" arm.
Arm/Group | Conventional Measures Only First; Then Conventional Measures + Hearing Aid | Conventional Measures + Hearing Aid First; Then Conventional Measures Only
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-06-01): https://cdn.clinicaltrials.gov/large-docs/24/NCT02269124/Prot_SAP_000.pdf
  • Informed Consent Form (2019-08-28): https://cdn.clinicaltrials.gov/large-docs/24/NCT02269124/ICF_001.pdf